CLINICAL TRIAL: NCT03285152
Title: A Feasibility Study Evaluating Metabolomic and Tissue Effects of Ketogenic Diet in Newly Diagnosed Overweight or Obese Endometrial Cancer Patients
Brief Title: A Study of Ketogenic Diet in Newly Diagnosed Overweight or Obese Endometrial Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-396
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer
Keywords: Ketogenic Diet; 17-396
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: This is a prospective, MSK investigator-initiated, multi-center, randomized, pilot study of KD vs SD consumption in treatment naïve endometrial cancer patients during the presurgical window period between diagnosis and surgical staging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (KD) (Experimental): The KD cohort will receive a rotating 7 day meal plan prepared by the Clinical Translational Science Center (CTSC) at Weill Cornell Medical Center (WCMC) with weekly food pick-up. The meal plan will provide a 3:1 fat to net carbohydrate ratio and calories for weight maintenance (30kcals /kg for a BMI< 30kg/ m2 and 25 kcal/kg for a BMI.30 kg/ m2.
  Interventions: Other: Ketogenic Diet (KD)
- Standard Diet (SD) (Active Comparator): Patients randomized to the SD group will consume their normal diet plan. They will meet with the dietitian from the CTSC at WCMC weekly and receive standard nutritional counseling from the CTSC. Average intake will be documented through analyzing a 3 day intake pre and post the 4 week period.
  Interventions: Other: Standard Diet (SD)

INTERVENTIONS:
Other: Ketogenic Diet (KD) — specially-formulated very low carbohydrate meals (KD)
  Arms: Ketogenic Diet (KD)
Other: Standard Diet (SD) — counseling on maintaining adequate nutritional intake from a normal diet (SD)
  Arms: Standard Diet (SD)

SUMMARY:
The purpose of this study is to test any good and bad effects of an experimental diet, called a ketogenic diet, in endometrial cancer. A ketogenic diet is one that is very low in carbohydrates (simple and complex sugars). The goal of this diet is for the body to go into a state of ketosis. Ketosis is when the body does not have enough sugar for energy so it burns stored fats which create acids called ketones, which can be used for energy. Researchers hope to learn whether or not a ketogenic diet is well-tolerated and safe to eat before surgery in endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis endometrial carcinoma on a tissue sample obtained at MSK (biopsy). Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, transitional cell carcinoma, carcinosarcoma.
* Age ≥ 18 years
* Patients must have consented to surgery with a board-certified Gyn surgeon
* Patients must have no had adjuvant therapy for the management of endometrial carcinoma. This includes chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen. This also pertains to hormonal, vascular, and targeted therapy for the management of endometrial cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with stage I-IVA are eligible
* Adequate hematologic defined by the following laboratory results obtained within 11 days prior to first study treatment:

  * Absolute neutrophil count (ANC) ≥1.5 k/mcl
  * Platelet count ≥ 100k/mcl
  * Hemoglobin ≥ 9.0 g/dL
* Adequate hepatic function defined by the following laboratory results obtained within 11 days prior to first study treatment:

  * Total bilirubin≤1.5x the upper limit of normal (ULN)
  * AST and ALT ≤ 3.0x ULN
  * Albumin ≥ 3.5 g/dL
* Adequate renal function defined by the following laboratory results obtained within 11 days prior to first study treatment:

  ° Serum creatinine≤1.5x ULN OR creatinine clearance ≥50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation
* HbA1c ≤ 7.9 %
* BMI ≥ 23 kg/m2
* Patients must agree to consent to the companion genomic profiling study MSK IRB# 12-245
* Patients must agree to consent for their tumor samples to be used for generation of cellular research tools such as organoids
* Willingness to travel to the CTSC at WCMC weekly
* Patient and/or Legally Authorized Representative must have the ability to read, write, speak and understand English. Note: If patient does not have the capability to read or write in English, the patient"s preferred language should be English and the LAR will be responsible for completing all study forms on the patient's behalf.

Exclusion Criteria:

* History of diabetes and on active diabetes treatment with pharmacotherapy (oral hypoglycemics or insulin)
* History of gout.
* History of myocardial infarction or unstable angina within 6 months prior to first study treatment.
* Active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection)
* New York Heart Association Class II or greater congestive heart failure.
* Patients with a QTc interval of >450 msec on screening electrocardiogram (ECG) for men or >470 msec for women.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption.
* Inability or unwillingness to swallow
* Clinically significant history of liver disease, including cirrhosis and current alcohol abuse.
* Known active hepatitis infection
* Known HIV infection.
* Need for current chronic corticosteroid therapy (≥ 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids)
* Pregnancy, lactation, or breastfeeding
* Patients of childbearing potential must have a negative pregnancy test within 11 days prior to treatment start to be eligible
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment.
* Known untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria:

  * Presence of measurable disease outside the CNS
  * No radiographic evidence of worsening upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
  * No history of intracranial hemorrhage or spinal cord hemorrhage
  * No ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
  * Absence of leptomeningeal disease
* Inability to comply with study and follow-up procedures
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* History of nephrolithiasis or nephrolithiasis including that incidentally discovered during CT screening.
* Known selenium deficiency
* Diagnosis of seizure disorder
* Participation in a diet (Atkins, Weight Watchers, Best Life, Nutrisystem, South Beach, Jenny Craig, Paleo Diet, Zone etc) or weight loss plan within 28 days prior to Day 1 of treatment that the investigator and/or nutritionist believes will confound results.
* Severe constipation or condition where exacerbation of constipation is not advisable (e.g. small bowel obstruction history)
* Planned vacation or dental work during the study phase that the investigator and/or nutritionist believes will impede the study plan
* Vegetarian or Vegan eating habits that cannot be accommodated by the nutrition team
* Untreated or poorly controlled gastro-esophageal reflux disease.
* An allergy or intolerance to egg, gluten or milk protein that cannot be accommodated by the nutrition team

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer Patients
Enrollment: 19 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
number of patients that complete the study | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Makker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent and Follow up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent & Follow Up), Harrison, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Rockville Centre, New York

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm